CLINICAL TRIAL: NCT06228079
Title: Adjuvant Therapy Versus Endoscopic Surgery Alone in Early-stage Recurrent Nasopharyngeal Carcinoma: A Multicenter Randomized Controlled Trial
Brief Title: Adjuvant vs Surgery Only in Early-stage Recurrent NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai 6th People's Hospital (Other); Changhai Hospital (Other); Fujian Medical University Union Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: early-rNPC-RCT-adj
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Immunotherapy; toripalimab; Drug Therapy; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The control group (No Intervention): Patients in the control group would go through observation and follow-up after recurrent endoscopic surgery.
- The experimental group (Experimental): Patients in the experimental group would be implemented with adjuvant therapy including chemotherapy and immunotherapy after endoscopic surgery.
  Interventions: Drug: Immunotherapy,Toripalimab Injection; Drug: Chemotherapy,Gemcitabine based regimen

INTERVENTIONS:
Drug: Immunotherapy,Toripalimab Injection — Patients in the experimental group would be implemented with adjuvant Immunotherapy and chemotherapy after endoscopic surgery. Four to six cycles chemotherapy and 10 cycles immunotherapy,or until unacceptable side effects.
  Arms: The experimental group
Drug: Chemotherapy,Gemcitabine based regimen — Patients in the experimental group would be implemented with adjuvant Immunotherapy and chemotherapy after endoscopic surgery. Four to six cycles chemotherapy and 10 cycles immunotherapy,or until unacceptable side effects.
  Arms: The experimental group

SUMMARY:
Adjuvant Therapy Versus Endoscopic Surgery Alone in Early-stage Recurrent Nasopharyngeal Carcinoma: A Multicenter Randomized Controlled Trial

DETAILED DESCRIPTION:
This study is an open-label, multicentered, evaluator-blinded , randomized clinical trial.

Patients with early-stage recurrent nasopharyngeal carcinoma were randomized into the control group and the experimental group. Patients in the control group would go through observation and follow-up after recurrent endoscopic surgery, while patients in the experimental group would be treated with adjuvant therapy such as chemotherapy and immunotherapy. A total of 176 subjects are required, with 88 patients in the control group and 88 patients in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with recurrent nasopharyngeal carcinoma;
2. Stage rT1 or rT2(superficial parapharyngeal space, distance to internal carotid artery >5mm)or rT3 (confined to the bottom wall of the sphenoid sinus),according to AJCC 8th edition;
3. Cervical lymph node metastasis can be controlled locally
4. Age 18 to 75 years;
5. Without distant metastasis;
6. Informed consent forms signed;
7. ≥6months from the accomplishment of radiation to recurrence
8. previously radiotherapy for only 1 course;
9. ECOG score 0-2 and can tolerate chemotherapy and immunotherapy
10. Sufficient organ function;
11. Undergone endoscopic surgery with negative pathological margin;

Exclusion Criteria:

1. Participation in other interventional clinical trials;
2. Uncontrolled illnesses which will interfere with the ability to undergo therapy;
3. Suffering from another or multiple malignancy within 5 years (excluding fully treated basal cell or skin squamous cell carcinoma, cervical carcinoma in situ);
4. Any contradiction to immune and chemotherapy;
5. With serious autoimmune disease;
6. Currently usage of immunosuppressive agents or systemic glucocorticoid therapy (dosage>10mg/day prednisone or other glucocorticoids), and continuing to use them within 2 weeks before the first administration of trial drugs;
7. Severe allergic reactions to other monoclonal antibodies;
8. History of radioactive particle planting;
9. Vaccination with live vaccine within 4 weeks prior to initial administration or possibly during the study period;
10. Female patients who are at pregnancy or lactation;
11. Other situations that the researchers believe are not suitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
DFS | From date of randomization until the date of first documented recurrence, metastasis or date of death from any cause, whichever came first, assessed up to 24 months
  Disease free survival

SECONDARY OUTCOMES:
OS | From randomization to death of any cause,assessed up to 60 months
  Overall Survival
LRFS | From randomization to local recurrence or death,assessed up to 24 months
  Local recurrence free survival
DMFS | From randomization to distant metastasis or death, assessed up to 24 months
  Distant metastasis free survival
1-and 2-year DFS rate | end of 1st year, end of 2nd year
  one- and two-year disease free survival
1-and 2-year OS rate | end of 1st year, end of 2nd year
  one- and two-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, Principal Investigator — Eye& ENT Hospital, Fudan University
Locations (7):
- China (7):
  - Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Fujian Medical University Union Hospital, Fuzhou
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Changhai Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shenzhen Second People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR